CLINICAL TRIAL: NCT02859766
Title: Evaluation of Safety and Systemic Pharmacokinetics After Single and Repeat Doses of Abicipar Pegol (AGN-150998) Intravitreal Injections in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Safety and Pharmacokinetics of Abicipar Pegol Intravitreal Injections in Patients With Neovascular AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150998-012
Record Dates: First submitted 2016-07-12; First posted 2016-08-09 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — abicipar pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abicipar Pegol_Repeat Dose (Experimental): Treatment Group 1: Abicipar pegol 2 mg administered to the study eye by intravitreal injection, 3 injections 4 weeks apart. [Day 1, Weeks 4 and 8]
  Interventions: Drug: Abicipar pegol
- Abicipar Pegol_Single Dose (Experimental): Treatment Group 2: Abicipar pegol 2 mg administered to the study eye by intravitreal injection on Day 1.
  Interventions: Drug: Abicipar pegol

INTERVENTIONS:
Drug: Abicipar pegol — Abicipar pegol 2 mg administered to the study eye by intravitreal injection.
  Other Names: AGN-150998

SUMMARY:
This study will evaluate the safety and characterize the systemic pharmacokinetics (PK) of free and vascular endothelial growth factor (VEGF)-bound abicipar following single and multiple intravitreal injections of abicipar pegol in treatment-naïve patients with neovascular age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

-Presence of active subfoveal and/or juxtafoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD).

Exclusion Criteria:

* History of or active periocular, ocular, or intraocular infection.
* Previous use of verteporfin photodynamic therapy (PDT) or any ocular anti-angiogenic therapy (eg, aflibercept, bevacizumab, ranibizumab, pegaptanib), approved or investigational, for the treatment of neovascular AMD or previous therapeutic radiation in the region.
* Prior use of ocular anti-VEGF agents for neovascular eye diseases other than AMD.
* Macular hemorrhage that involves the center of fovea in the study eye.
* Any prior or current systemic or ocular treatment (including surgery) for neovascular AMD in the study eye.
* Treatment with ocular corticosteroid injections or implants within 6 months in the study eye.
* History or evidence of eye surgery: Pars plana vitrectomy, Submacular surgery or other surgical interventions for AMD, Incisional glaucoma surgery or Cataract or refractive surgery within the last 3 months.
* AMD in the non-study eye that requires anti-VEGF treatment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Peak Serum Concentration (CMax) for Free and VEGF-Bound Abicipar | Treatment Group 1: Baseline to Week 20 and Treatment Group 2: Baseline to Week 12
Serum Concentration Immediately before Next Dose (Ctrough) for Free and VEGF-Bound Abicipar | Treatment Group 1: Baseline to Week 20 and Treatment Group 2: Baseline to Week 12
Time to Cmax (Tmax) for Free and VEGF-Bound Abicipar | Treatment Group 1: Baseline to Week 20 and Treatment Group 2: Baseline to Week 12
Terminal Elimination Half-Life (t1/2) for Free and VEGF-Bound Abicipar | Treatment Group 1: Baseline to Week 20 and Treatment Group 2: Baseline to Week 12
Area Under the Serum Concentration-Time Curve from Zero to the End of the Dosing Interval "tau" (AUC0-tau) for Free and VEGF-Bound Abicipar | Treatment Group 1: Baseline to Week 20 and Treatment Group 2: Baseline to Week 12
Area Under the Serum Concentration-Time Curve from Zero to Infinity (AUC0-inf) for Free and VEGF-Bound Abicipar | Treatment Group 1: Baseline to Week 20 and Treatment Group 2: Baseline to Week 12

SECONDARY OUTCOMES:
Serum Levels of Anti-abicipar Antibodies | Treatment Group 1: Baseline to Week 20 and Treatment Group 2: Baseline to Week 12
Percentage of Participants with Treatment Emergent Adverse Events | Treatment Group 1: Baseline to Week 20 and Treatment Group 2: Baseline to Week 12
Best Corrected Visual Acuity using an Eye Chart | Treatment Group 1: Baseline to Week 20 and Treatment Group 2: Baseline to Week 12
Percentage of Participants with Change from Baseline in Full Ophthalmic Exam Findings [i.e. Slit Lamp Exam, Intraocular Pressure (IOP) Measurements, Funduscopic Exam] | Treatment Group 1: Baseline, Week 20 and Treatment Group 2: Baseline, Week 12
Changes from Baseline in General Physical Condition as Measured through General Physical Exam | Treatment Group 1: Baseline, Week 20 and Treatment Group 2: Baseline, Week 12
Percentage of Participants with Changes from Baseline in Vital Signs (Blood Pressure, Pulse Rate) | Treatment Group 1: Baseline, Week 20 and Treatment Group 2: Baseline, Week 12
Percentage of Participants with Change from Baseline in Clinically Relevant Laboratory Values (Serum Chemistry, Hematology, Urinalysis) | Treatment Group 1: Baseline, Week 20 and Treatment Group 2: Baseline, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Sutherland, Study Director — Allergan
Locations (18):
- United States (18):
  - Retinal Consultants of Arizona, Gilbert, Arizona
  - Win Retina, Arcadia, California
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Atlantis Retina Institute (Atlantis Eyecare), Huntington Beach, California
  - Jacobs Retina Center, Shiley Eye Institute, UCSD, La Jolla, California
  - California Eye Specialists Medical Group, Inc-Private Clinic, Pasadena, California
  - University of Miami, Coral Gables, Florida
  - The Eye Institute of West Florida, Largo, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - East Florida Eye Insititute, Stuart, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Raj K. Maturi, MD, Indianapolis, Indiana
  - Massachusetts Eye & Ear, Boston, Massachusetts
  - Eyesight Ophthalmic Services, PA, Portsmouth, New Hampshire
  - Caroline Eye Associates, Southern Pines, North Carolina
  - Cole Eye Institute, Cleveland Clinic, Cleveland, Ohio
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - Davis Duehr Dean, Madison, Wisconsin